CLINICAL TRIAL: NCT04664530
Title: The Study on the Esketamine in the Treatment of Postherpetic Neuralgia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-1035
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Postherpetic Neuralgia; Esketamine
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Esketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Drug: Saline
- Treatment group (Experimental)
  Interventions: Drug: esketamine

INTERVENTIONS:
Drug: esketamine — The in-hospital intervention process is divided into a titration phase and an effect evaluation phase. After admission, all patients received pregabalin 150mg twice for one day and amitriptyline 12.5mg one piece per night. The treatment group was combined with intranasal esketamine three times per day, and individualized concentration titration was performed within 5 days. Set the initial dosage to 10mg for nasal drops. If the score is less than 5 points compared to the basic value, the dose is increased by 5 mg each time. When the dose reaches 25mg, the increment of the dose will be adjusted to 10mg. If the score is reduced by ≥5 points compared to the basic value, the current dose will be maintained and the titration will end. The titration phase will be finished when the titration dose reaches 35mg or untolerable adverse reactions occurs. Finally, a 7 tesla scan was performed on the right-hand patients with herpes on the body to explore the effect of ketamine on the brain network.
  Arms: Treatment group
Drug: Saline — The titration process in the control group with saline are the same as those in the treatment group with esketamine.
  Arms: Control group

SUMMARY:
Herpes zoster (HZ) is an acute herpetic skin disease caused by the reactivation of the varicella-zoster virus (VZV) latent in the sensory ganglia. Postherpetic neuralgia (PHN) often occurs after herpes zoster heals and persists for a long time. At present, clinically anticonvulsants (such as gabapentin, pregabalin) and antidepressants (such as amitriptyline) are clinically first-line drugs for the treatment of PHN, which are not usually effective to treat PHN well, as well as to alleviate patients' bad mental symptoms. Esketamine, as a well-known N-methyl-D-aspartate receptor inhibitor, has both analgesic and antidepressant effects with extremely few incidence of respiratory depression, delirium, hallucinations, nausea and vomiting. Therefore, we hypothesize that esketamine could relieve PHN and Anxiety and depression-like symptoms symptoms in patients with PHN. This study intended to compare the efficacy of pregabalin, amitriptyline combined with esketamine therapy and pregabalin combined with amitriptyline therapy for alleviating PHN, and to further explore the feasibility and safety of esketamine in the treatment of PHN as well as underlying the mechanism of esketamine on the PHN.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old; Patients with post-herpetic neuralgia with anxiety and depression; NRS ≧4 points; A and (or) D ≧8 points in the Hospital Anxiety and Depression Scale (HADS) ; The course of disease ≧3 months; Patients with invalid conventional treatment (pregabalin or gabapentin combined with anti-anxiety depression, anti-epileptic dugs).

Exclusion Criteria:

* Present acute and chronic pain caused by other disease during treatment; Serious systemic disease; Severe infection, history of heart, lung, liver and kidney dysfunction, tumor, immunodeficiency and other serious diseases, or currently receiving or have recently received immunosuppression or cytotoxic drug treatment; A history of mental illness such as epilepsy, depression, Alzheimer's, multiple sclerosis, Parkinson, etc., and a history of head trauma; Participating in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scales | Baseline, once for the period of drug administration
  The score to assess the pain degree

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Study Chair — The second affiliated hospital of Zhejiang University hangzhou, Zhejiang, China
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided